CLINICAL TRIAL: NCT00650338
Title: A Randomized, Double-masked, Placebo- and Active- Controlled, Parallel-group, Multi-center, Dose-response Trial of DE-104 Ophthalmic Solution in Subjects With Primary Open-angle Glaucoma or Ocular Hypertension
Brief Title: Safety and Efficacy Study of DE-104 Ophthalmic Solution to Treat Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27-002
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Experimental): <described in intervention>
  Interventions: Drug: DE-104 ophthalmic solution, low concentration
- 2 (Experimental): <described in intervention>
  Interventions: Drug: DE-104 ophthalmic solution, medium concentration
- 3 (Experimental): <described in intervention>
  Interventions: Drug: DE-104 ophthalmic solution, high concentration
- 4 (Placebo Comparator): <described in intervention>
  Interventions: Drug: Placebo
- 5 (Active Comparator): <described intervention>
  Interventions: Drug: 0.005% latanoprost

INTERVENTIONS:
Drug: DE-104 ophthalmic solution, low concentration — Topical ocular application
  Arms: 1
Drug: DE-104 ophthalmic solution, medium concentration — Topical ocular application
  Arms: 2
Drug: DE-104 ophthalmic solution, high concentration — Topical ocular application
  Arms: 3
Drug: Placebo — placebo
  Arms: 4
Drug: 0.005% latanoprost — Topical ocular application
  Arms: 5

SUMMARY:
To investigate the dose-response relationship of DE-104 ophthalmic solution in lowering intraocular pressure (IOP) in subjects with Primary Open-Angle Glaucoma or Ocular Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Provided signed, written informed consent.
* Diagnosed with primary open-angle glaucoma or ocular hypertension.
* 18 years of age and older.
* If a subject is a female of childbearing potential, she must utilize reliable contraceptive throughout the study, and must have a negative urine pregnancy test prior to enrollment into this study.

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy, or females of childbearing potential who are not using a reliable method of contraception.
* Presence of any abnormality or significant illness that could be expected to interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To investigate the dose-response relationship of DE-104 in lowering intraocular pressure (IOP) | 28 days

SECONDARY OUTCOMES:
To compare the safety and efficacy of DE-104 ophthalmic solution with placebo and 0.005% latanoprost. | 35 days

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Sall Research Medical Center, Artesia, California
  - USC Department of Ophthalmology, Los Angeles, California
  - Wolstan Eye Associates, Torrance, California
  - East Florida Eye Institute, Stuart, Florida
  - Seidenberg Protzko Eye Associates, Bel Air, Maryland
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Cornerstone Eye Care, High Point, North Carolina
  - Associated Glaucoma Consultants, Philadelphia, Pennsylvania
  - Keystone Research, Ltd., Austin, Texas
  - David Shulman, MD P-A, San Antonio, Texas
  - Eye Clinics of South Texas, San Antonio, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Virginia Eye Consultants, Norfolk, Virginia